CLINICAL TRIAL: NCT04812626
Title: Efficacy and Safety of Intralesional Triamcinolone Acetonide Alone and Its Combination With 5-fluorouracil in Keloids and Hypertrophic Scars
Brief Title: Intralesional Triamcinolone Acetonide and Its Combination With 5-fluorouracil in Keloids and Hypertrophic Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Collaborators: Nepal Health Research Council (Other Government)
Responsible Party: Principal Investigator, Ripala Acharya, Junior resident, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BPK
Record Dates: First submitted 2021-03-06; First posted 2021-03-23 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2021-03

CONDITIONS: Scar Keloid
MeSH Terms: conditions — Keloid | interventions — Fluorouracil; Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel Group, Double Blinded, Clinical Trial Group A: Will receive Intralesional Triamcinolone acetonide only Group B: Will receive Intralesional Triamcinolone acetonide + 5 fluorouracil combination
Who Masked: Participant, Care Provider
Masking Description: This study will be double blinded with both the participants (keloid/hypertrophic scar patient fulfilling all the criteria)) and trial investigator (treatment provider) being blinded. The participants will be unaware of the treatment group that they will be allocated. And even the investigator performing the procedure and assessing the scar in each visit will be unaware of the drugs that will be given.
  The independent dermatologist, which will have the sealed envelope will open the envelope and instruct the trained nurse to prepare the mixture of drugs as the group written in the envelope and provide it to the blinded investigator after removing the label on the mixture of drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Intralesional (IL) triamcinolone acetonide (TAC) alone; (Experimental): Group A: 1 ml of 40mg/ml triamcinolone acetonide will be mixed with 1ml of normal saline. 5 units (0.125ml) of the mixture will be given intralesional with the help of 1ml insulin syringe of 40units,covering an area of 0.5X0.5 cm2 of scar. Each extra area of 0.5x0.5cm2 will be given 5 units of injection of above mixture of drugs( maximum dose=2ml). Follow up Injection will be given at 2 weeks interval for total of 6 sessions (at 0,2, 4, 6,8,10 weeks) Post treatment follow up: at 12 weeks.
  Interventions: Drug: 5-Fluorouracil
- Group B: Intralesional triamcinolone acetonide and 5-fluorouracil (5-FU) combination (Experimental): Group B: 1 ml of 40 mg/ml triamcinolone acetonide will be mixed with 1ml of 50 mg/ml FU.
  Injection Method: Five units (0.125ml) of the mixture will be given intralesional with the help of 1ml insulin syringe of 40units, that covers an area of about 0.5X0.5 cm2 of scar, each extra area of 0.5x0.5cm2 will be given 5 units of injection of above mixture of drugs. (maximum dose 2ml). Follow up Injection will be given at 2 weeks interval for total of 6 sessions (at 0,2, 4, 6,8,10 weeks), Post treatment follow up: at 12 weeks.
  Interventions: Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: 5-Fluorouracil — Group A: 1ml of 40mg/ml triamcinolone acetonide will be mixed with 1ml of normal saline Group B:1 ml of 40 mg/ml triamcinolone acetonide will be mixed with 1ml of 50 mg/ml FU Five units (0.125ml) of the mixture TAC 40mg/ml and 5-FU 50mg/ml (1:1) i.e. 2.5mg TAC and 3.125mg of 5-FU or TAC 40mg/ml and 2%xylocaine (1:1) i.e. 2.5mg of TAC will be given intralesional with the help of 1ml insulin syringe of 40units, that covers an area of about 0.5X0.5 cm2 of scar, thus, a scar of 1 cm2 will require 4 injections to cover the whole lesion. Each extra area of 0.5x0.5cm2 will be given 5 units of injection of above mixture of drugs. For the larger lesions, dose can be increased but no more than 2ml in each group. Injection will be given at 2 weeks interval for total of 6 sessions (at 0,2, 4, 6,8,10 weeks) Post treatment follow up: at 12 weeks.
  Other Names: Triamcinolone acetonide

SUMMARY:
Summary: Keloids and hypertrophic scars are benign fibrous growth, differing mainly by overgrowth beyond the initial defect in keloid whereas hypertrophic scar is confined to initial lesion and tends to regress over the years. Keloids and hypertrophic scars mainly lead to cosmetic disfigurement and functional deformity depending on site of involvement, in addition to symptoms like pain and pruritus, encountered occasionally. These sometimes might lead to psychological impact too. Different treatment options for keloids and hypertrophic scar are silicone gel/ sheets, corticosteroids, cryotherapy, lasers, antineoplastic agents (5-FU, mitomycin-C), surgical excision and immunomodulators (imiquimod) used either as monotherapy or combination therapy. Different studies involving combination of TAC and 5-FU have been done so far which shows better treatment outcome in terms of efficacy and safety. In a recent meta-analysis published in 2017 concluded that combination therapy of 5-FU + TAC offers better outcome than TAC alone, however recommended additional randomized, controlled, large-sample, high quality trial are needed for a more objective analysis of the treatment efficacy and to assess the adverse reaction associated. We are conducting this study the objective to compare the efficacy and safety profile of intralesional triamcinolone acetonide alone and its combination with 5-FU of the treatment of keloids and hypertrophic scars. This study may help in finding out the optimum treatment option in keloid and hypertrophic scar with minimal side effects in our clinical practice.

DETAILED DESCRIPTION:
HYPOTHESIS Null hypothesis: There is no difference in the efficacy of intralesional triamcinolone acetonide alone and its combination with 5-flurouracil in the treatment of keloids and hypertrophic scars Alternate hypothesis: Combination of intralesional triamcinolone and 5- fluorouracil is more efficacious than intralesional triamcinolone alone in treatment of keloids and hypertrophic scars

METHODS

Sample size: Sample size:

This study considers a 95% confidence interval, 80% power to estimate sample size. According to the article published in the Clinical and experimental dermatology by Darougegh A et al in 2009 comparing the efficacy of Intralesional Triamcinolone alone versus combined with 5 FU in treatment of keloids, it was found that the patient reported good to excellent (> 50%) 30 | P a g e improvement in TAC alone group was 20% whereas that of the combination of TAC and 5-FU was 55% (22). Now using the sample size estimation formula for 2 proportions based on above study, n = {2p(1-p) (Zβ + Zα/2)2}/ (p1-p2)2 Where n= sample size for each group; p1 = 0.55; p2 = 0.2; p= (p1 +p2)/2; Zα/2=1.96 at 95% CI; Zβ = 0.842 at 80% power; using above formula, n= 30. Adding 10% in calculated value to consider the drop out, the minimum sample size in each group will be 30+3=33; Thus, a total sample size will be 66 The study is double blinded ,both participants and investigator( treatment provider/assessor) are blinded. Total of 66 patients are enrolled into the study , 33 in each groups allocated by block randomization through computer generated block randomization list. Patients with a clinical diagnosis of keloids or hypertrophic scars attending the outpatient department of dermatology at BPKIHS will be enrolled in the study. Written and understood informed consent will be taken prior to the enrollment and treatment. Detailed information of all the patients satisfying inclusion criteria will be recorded in preset pro forma. This will include personal data, past history, medical history, drug history, clinical data like site, size, number, distribution of lesions, complaints related to scar like pain, pruritus, erythema, scar score and cutaneous examination. Patients will be excluded according to the exclusion criteria. Photographs of the lesions will be taken before the first treatment session, in every treatment session and at the completion of treatment at 12th week. Only one lesion (preferably on the trunk or proximal extremity) will be treated per patient.

Study Treatments:

Each patient will be assigned a patient identity number and will be allocated to receive either triamcinolone acetonide alone (1ml of 40mg/ml triamcinolone acetonide will be mixed with 1ml of normal saline) or triamcinolone acetonide and 5-FU combination (1ml of 40 mg/ml triamcinolone acetonide will be mixed with 1ml of 50 mg/ml FU) depending upon the treatment specified in the sealed opaque envelope.

Treatment will be provided as follows:

Group A: Intralesional Triamcinolone only One ml of 40mg/ml triamcinolone acetonide will be mixed with 1ml of normal saline to make a 20mg/ml concentration.

Group B Intralesional Triamcinolone + 5 fluorouracil One ml of 40 mg/ml triamcinolone acetonide will be mixed with 1ml of 50 mg/ml FU with resulting mixture TAC/5-FU concentration being 20mg/25mg per ml .

Treatment duration: 10 weeks (drug given at 0,2, 4, 6,8,10 weeks)

Post treatment follow up: at 12 weeks.

Assessment:

During treatment and during follow-ups, the scar will be assessed for the following:

1. Length, width and height of the scar: using Vernier calipers and digital photography
2. POSAS scoring:
3. Vancouver Scar Scale (VSS)
4. Subjective improvement: Overall improvement as graded by patient and observer separately on a 5 point scale and percentage in improvement is assessed in each follow up visit (no/poor: up to 25% , fair: 26-50%, good: 51-75%, excellent : 76-100% improvement) and efficacy is determined by good to excellent improvement( improvement >50%) in patient and observer reported separately

Efficacy evaluation:

The primary efficacy endpoints will be calculated on the basis of the percent reduction from baseline to week 12 in the subjective improvement, lesion size and scar scores and taking single lesion as the reference lesion in a patient (in case of multiple number of lesions under treatment in a single patient). The response rates (percentage of patients achieving 50% reduction in size of scar, percentage of patient achieving good to excellent subjective improvement) will also be compared at 12 weeks in each treatment group.

Safety evaluation: Safety of treatment is assessed through evaluation of local adverse effects like erythema, pain, atrophy, ulceration, telangiectasia, pigmentation and systemic effects if any like Cushing's syndrome in each follow up visit week 2, 4, 6, 8, 10 and 12.

Statistical analysis Data will be entered in Microsoft Excel 2016 (Microsoft Corporation, Redmond, Washington, USA) and statistical analysis will be done using Statistical Package for the Social Sciences 11.5 version (Chicago, Inc). Statistical analysis will be conducted both per-protocol and intention-to treat population (defined as all enrolled patients to whom study drug will be given; with the last observation carried forward) basis using two sided tests.

For descriptive statistics, percentage, mean, Standard Deviation, median, interquartile range and minimum, maximum will be calculated along with graphical and tabular presentation. For inferential statistics, statistical methods proposed are as follow Chi square test , Paired t test ,Independent 't' test ,Wilcoxon signed rank test , Mann- Whitney U test , Kaplan-Meier curves The test of significance will be considered when the value of p< 0.05

ELIGIBILITY:
Inclusion Criteria:

1. Patient with clinically diagnosed keloid or hypertrophic scar
2. Size of scar 1cm in length or more
3. Informed consent given

Exclusion Criteria:

1. Under treatment of keloids or hypertrophic scar in past 6 months
2. Patient with renal disease
3. Patient with liver disease
4. History of Hypersensitivity to 5-fluorouracil or triamcinolone acetonide
5. Immunosuppressed conditions: HIV, Immunosuppressive therapy, Uncontrolled diabetes
6. Pregnant or lactating women or patient planning for pregnancy
7. Open wound in the scar
8. Atrophic scar
9. Patients suffering from chronic infectious conditions like Tuberculosis
10. Patients with low WBC count

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-08-14 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Percentage of change in height of scar pre and post treatment in each groups | Starting of treatment to 12 weeks follow up of treatment
  Compare the change in height in millimeter of scar pre and post treatment in percentages in each treatment groups
Percentage of reduction in The Patient and Observer Scar Assessment Score) score in two treatment groups | Starting of treatment to 12 weeks follow up of treatment
  Compare the reduction in The Patient and Observer Scar Assessment Score from baseline to 12 week follow up in each group in percentage
Percentage of change in Vancouver Scar Scale score in two treatment groups | Starting of treatment to 12 weeks follow up of treatment
  Compare the change in Vancouver Scar Scale from baseline to 12 week follow up in each group in percentage
Percentage of good to excellent subjective improvement in two groups combination with 5-flurouracil in the treatment of keloids and hypertrophic scars at 12 weeks follow up | Starting of treatment to 12 weeks follow up of treatment
  Compare the good to excellent improvement (>50% subjective improvement) in the scars in two treatment groups in percentage

SECONDARY OUTCOMES:
Percentages of Side effects of treatment groups | Starting of treatment to 12 weeks follow up of treatment
  Compare the percentages of side effects of treatment between the group

CONTACTS AND LOCATIONS:
Overall Officials: Ripala Acharya, MBBS, Principal Investigator — B.P. Koirala Institute of Health Sciences
Locations (1):
- B.P. Koirala Institute of Health Sciences, Dharān, Province No. 1, Nepal

IPD SHARING:
Plan to Share IPD: No